CLINICAL TRIAL: NCT04190615
Title: Determination of Reference Ranges of Thromboelastometry ClotPro Analyser in Paediatric Patients Undergoing Elective Surgery
Brief Title: Determination of ClotPro Paediatric Reference Range Study
Status: Completed | Type: Observational
Sponsor: National Institute of Children's Diseases, Slovakia (Other Government)
Responsible Party: Principal Investigator, Katarina Laukova, MD, Paediatric Anaesthetist, Attending physician, National Institute of Children's Diseases, Slovakia
Other Study IDs: NICDOS1TEMCP
Record Dates: First submitted 2019-11-30; First posted 2019-12-09 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Clotting and Bleeding Disorders; Child Development; Infant Development; Coagulopathy
Keywords: thromboelastometry; viscoelastic testing; reference ranges
MeSH Terms: conditions — Thrombosis; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 0 to 3 months: 0 (term newborns) to 3 month of age
  Interventions: Diagnostic Test: thromboelastometry test (TEM test)
- 4 to12 months: infants from 4month to 12month of age
  Interventions: Diagnostic Test: thromboelastometry test (TEM test)
- 13 to 24 months: children from 13month to 2years of age
  Interventions: Diagnostic Test: thromboelastometry test (TEM test)
- 2 to 5 years: children from 2 to 5 years of age
  Interventions: Diagnostic Test: thromboelastometry test (TEM test)
- 6 to 10 years: children from 2 to 10 years of age
  Interventions: Diagnostic Test: thromboelastometry test (TEM test)
- 11 to16 years: children from 11 to 16 years of age
  Interventions: Diagnostic Test: thromboelastometry test (TEM test)

INTERVENTIONS:
Diagnostic Test: thromboelastometry test (TEM test) — TEM test from the whole blood sample

SUMMARY:
A new thromboelastometry analyser (ClotPro, Enicor GmbH, Munich, Germany) with improved technology was developed. This device has an improved new-generation viscoelastometric testing technique and enables the detection and assessment of factor deficiencies, low fibrinogen, platelet contribution (to whole blood coagulation), heparin and direct oral anticoagulants effects, fibrinolysis and antifibrinolytic drugs. This study aims to determine reference ranges for the ClotPro device for all paediatric age groups.

DETAILED DESCRIPTION:
Viscoelastic testing as a relatively novel method to assess coagulation status appears favourable in reducing blood product transfusions. The tests are performed on whole blood instead of plasma, which saves time and gives a quick sight at the interaction between cellular and plasmatic clotting factors.

Reviews of the literature suggest that transfusions of packed red blood cells (pRBC), plasma, and platelets are all decreased in patients whose transfusions were guided by viscoelastic tests rather than by clinical judgement or conventional laboratory tests.

The benefits of viscoelastic coagulation monitoring have been described in many fields of surgery and intensive care. Current literature and a guideline for the treatment of massive haemorrhage in perioperative bleeding and trauma patients recommend the use of viscoelastic tests to guide haemostatic resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* paediatric patients attending hospital for elective surgery or diagnostic imaging undergoing general anaesthesia are going to be eligible to participate.
* children whose parents agree to participate are provided with oral and written information and written informed consent has to be obtained.

Exclusion Criteria:

* problematic blood collection
* age over 16 years
* emergency surgery
* systemic infection
* known bleeding disorders
* history of congenital or acquired coagulopathy including renal, liver and bone marrow disease,
* any medication interfering with haemostasis
* prophylactic or therapeutic anticoagulant therapy (acetylsalicylic acid within the last 10 days or low-molecular-weight heparins within the last 48 h)
* administration of colloids hydroxyethyl starch (HES)/albumin, or blood products before the blood withdrawal

Ages: 1 Hour to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 6 Individual age categories are determined to monitor: ASA physical status I-II
  1. 0 (full term) to 3 months
  2. 4 to12 months
  3. 13 to 24 months
  4. 2 to 5 years
  5. 6 to10 years
  6. 11 to 16 years Demographic data to be recorded: age, gender, weight, height.
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
reference range for the thromboelastometry analyser (ClotPro, Enicor GmbH, Munich, Germany) in age group 0 to 3 months for EX-test, FIB-test, IN-test, HI-test, RVV test and TPA test | 30 minutes post blood sampling
  Measurement of thromboelastometry parameters in paediatric patients of 0-3months age group undergoing elective surgery or diagnostic procedure requiring general anaesthesia.
reference range for the thromboelastometry analyser (ClotPro, Enicor GmbH, Munich, Germany) in age group 4 to 12 months for EX-test, FIB-test, IN-test, HI-test, RVV test and TPA test . | 30 minutes post blood sampling
  Measurement of thromboelastometry parameters in paediatric patients of 4-12months age group undergoing elective surgery or diagnostic procedure requiring general anaesthesia.
reference range for the thromboelastometry analyser (ClotPro, Enicor GmbH, Munich, Germany) in age group 13 to 24 months for EX-test, FIB-test, IN-test, HI-test, RVV test and TPA test . | 30 minutes post blood sampling
  Measurement of thromboelastometry parameters in paediatric patients of 13-24months age group undergoing elective surgery or diagnostic procedure requiring general anaesthesia.
reference range for the thromboelastometry analyser (ClotPro, Enicor GmbH, Munich, Germany) in age group 2 to 5 years for EX-test, FIB-test, IN-test, HI-test, RVV test and TPA test | 30 minutes post blood sampling
  Measurement of thromboelastometry parameters in paediatric patients of 2-5years age group undergoing elective surgery or diagnostic procedure requiring general anaesthesia.
reference range for the thromboelastometry analyser (ClotPro, Enicor GmbH, Munich, Germany) in age group 6 to10 years for EX-test, FIB-test, IN-test, HI-test, RVV test and TPA test | 30 minutes post blood sampling
  Measurement of thromboelastometry parameters in paediatric patients of 6 to10 years group undergoing elective surgery or diagnostic procedure requiring general anaesthesia.
reference range for the thromboelastometry analyser (ClotPro, Enicor GmbH, Munich, Germany) in age group 11-16 years for EX-test, FIB-test, IN-test, HI-test, RVV test and TPA test | 30 minutes post blood sampling
  Measurement of thromboelastometry parameters in paediatric patients of 11-16 years group undergoing elective surgery or diagnostic procedure requiring general anaesthesia.

SECONDARY OUTCOMES:
Age related differences in thromboelastometry parameters | 12 months
  possible differences in monitored parameters across age groups;
Gender-related differences in thromboelastometry parameters | 12 months
  possible differences in parameters between genders.

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Laukova, MD, Principal Investigator — National Institute of Children's Diseases, Bratislava
Locations (1):
- National Institute of Children's Diseases, Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Laukova K, Petrikova V, Poloniova L, Babulicova L, Wsolova L, Haas T. Determination of reference ranges for the ClotPro(R) thromboelastometry device in paediatric patients. Br J Anaesth. 2023 Feb;130(2):183-190. doi: 10.1016/j.bja.2022.09.023. Epub 2022 Nov 12. PMID 36376099